CLINICAL TRIAL: NCT02873780
Title: Comparison of 3-Minute Step Test (3MStepT) and 6-Minute Walk Test (6MWT) in Chronic Obstructive Pulmonary Disease Patients
Brief Title: Comparison of 3-Minute Step Test (3MStepT) and 6-Minute Walk Test (6MWT) in COPD Patients
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier des Pays de Morlaix (Other)
Collaborators: Cliniques universitaires Saint-Luc- Université Catholique de Louvain (Other)
Responsible Party: Principal Investigator, Marc Beaumont, physiotherapist, Centre Hospitalier des Pays de Morlaix
Other Study IDs: BE403201317621
Record Dates: First submitted 2016-07-31; First posted 2016-08-22 (Estimated); Last update posted 2017-01-31 (Estimated); Status verified 2017-01

CONDITIONS: COPD; Chronic Obstructive Pulmonary Disease
Keywords: Pulmonary rehabilitation; COPD; Evaluation; oxygen desaturation; exercise capacity
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
The aim of this study is to compare oxygen desaturation during two tests: the 6 minute walk test and the 3 minute step test, for COPD patients.

DETAILED DESCRIPTION:
The 6 minute walk test (6MWT) is the best field test to determine oxygen desaturation during effort, in COPD patients. However, the test need a 30m corridor.

The 3 minute step test (3MST) is a other field test used in COPD patients. But no study shows that 3MST can be used to determine oxygen desaturation.

The aim of this study is to compare oxygen desaturation during these to tests : the 6MWT and the 3MST.

50 patients will be included in this study.

Patients realize two 6MWT and two 3MST, with rest between each test.

Oxygen saturation, heart rate are registered during the tests, dyspnea, leg peniblility are notified before and after each test, distance or number of steps are noted.

ELIGIBILITY:
Inclusion Criteria:

* stable COPD patients hospitalized for pulmonary rehabilitation program

Exclusion Criteria:

* acute exacerbation of COPD
* incapacity to realize the tests
* absence of written informed consent

Ages: 40 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: COPD patients hospitalized for pulmonary rehabilitation program
Sampling Method: Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2016-07; Primary Completion 2016-09 (Actual); Study Completion 2016-09 (Actual)

PRIMARY OUTCOMES:
oxygen saturation | 3 minutes
  oxygen saturation is compared between 6MWT and 3MST at the end of the 2 tests

SECONDARY OUTCOMES:
heart rate | 3 minutes
  heart rate is compared between 6MWT and 3MST at the end of the 2 tests
dyspnea (Borg Scale) | 3 minutes
  dyspnea (Borg Scale) is compared between 6MWT and 3MST at the end of the 2 tests
leg penibility (Borg Scale) | 3 minutes
  leg penibility (Borg Scale) is compared between 6MWT and 3MST at the end of the 2 tests

CONTACTS AND LOCATIONS:
Overall Officials: Marc Beaumont, PT, Principal Investigator — France, Britain, CH Des Pays de Morlaix; Gregory Reychler, PT, PhD, Principal Investigator — Belgium, Cliniques universitaires de Saint Luc
Locations (1):
- CH Des pays de Morlaix, Morlaix, France

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Result] Roberts MM, Cho JG, Sandoz JS, Wheatley JR. Oxygen desaturation and adverse events during 6-min walk testing in patients with COPD. Respirology. 2015 Apr;20(3):419-25. doi: 10.1111/resp.12471. Epub 2015 Jan 20. PMID 25601398
- [Result] Polkey MI, Spruit MA, Edwards LD, Watkins ML, Pinto-Plata V, Vestbo J, Calverley PM, Tal-Singer R, Agusti A, Bakke PS, Coxson HO, Lomas DA, MacNee W, Rennard S, Silverman EK, Miller BE, Crim C, Yates J, Wouters EF, Celli B; Evaluation of COPD Longitudinally to Identify Predictive Surrogate Endpoints (ECLIPSE) Study Investigators. Six-minute-walk test in chronic obstructive pulmonary disease: minimal clinically important difference for death or hospitalization. Am J Respir Crit Care Med. 2013 Feb 15;187(4):382-6. doi: 10.1164/rccm.201209-1596OC. Epub 2012 Dec 21. PMID 23262518
- [Result] Holland AE, Spruit MA, Troosters T, Puhan MA, Pepin V, Saey D, McCormack MC, Carlin BW, Sciurba FC, Pitta F, Wanger J, MacIntyre N, Kaminsky DA, Culver BH, Revill SM, Hernandes NA, Andrianopoulos V, Camillo CA, Mitchell KE, Lee AL, Hill CJ, Singh SJ. An official European Respiratory Society/American Thoracic Society technical standard: field walking tests in chronic respiratory disease. Eur Respir J. 2014 Dec;44(6):1428-46. doi: 10.1183/09031936.00150314. Epub 2014 Oct 30. PMID 25359355